CLINICAL TRIAL: NCT04163731
Title: VAlidation of an Self Administered Questionnaire in French for Assessment of Cardio Respiratory Reserve
Acronym: VAQAR
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0409; 2019-A02629-48 (Other: ID-RCB)
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stable patient, referred for a VO2 peak test: All stable patients above 18 years, referred for a VO2 peak test as part of their standard management in the Louis Pradel Hospital (Hospices Civils de Lyon, Lyon) and without acute clinical event in the last 3 months. All patients who accept to participate will undergo a self-questionnaire of 10 minutes.
  Interventions: Other: DASI questionnaire

INTERVENTIONS:
Other: DASI questionnaire — All patients who accept to participate will undergo a self-questionnaire of 10 minutes. Medical data of their cardiac stress test and risk factor will be collected.

SUMMARY:
The guidelines of the European Society of Cardiology (ESC) for preoperative management in non-cardiac surgery make the estimation of patients' maximum oxygen uptake (VO2peak) one of the cornerstones of preoperative evaluation.

Indeed, below a certain threshold of VO2 peak fixed in the literature at 15 milliliters/kilogram/minutes (ml/kg/min) (or 4 Metabolic Equivalent of Task - MET), the ESC recommends to carry out additional non-invasive examinations to evaluate the coronary risk of these patients.

In current practice, this evaluation is performed in anesthesia consultation by non-standard interview. The question "Can you go up a floor or climb a hill?" permits to classify patients with more or less VO2 peak than 4 MET.

However, several studies, including one published in the Lancet in 2018, show that this evaluation doesn't assess correctly the VO2peak of the patients nor predict post-operative cardiac complications.

In the same study, the evaluation of a standardized self-questionnaire, the Duke Activity Status Index (DASI), found a good correlation between the value of this pre-operative score and the 30-day mortality as well as the occurrence of infarction.

This self-questionnaire contains a dozen questions about the physical activities of daily life that patients are able or not to perform (household, various physical activity). It has also been validated in medical patients as being well correlated with the value of VO2 peak in the case of an answer by a third party (r = 0.81, p <0.001) and satisfactory in the case of a self-questionnaire (r = 0.58 , p <0.001).

This self-questionnaire exists in English but there is no validated translation in French. Given the cultural differences, it seems necessary in order to use it in a French-speaking context to go through a scientific validation stage. A validation study of DASI in Portuguese has already been published recently, serving as a methodological basis for a French translation.

The purpose of this study is to carry out a validation of a standardized self-questionnaire in French. It will be distributed to patients referred for a VO2peak test as part of their standard management in the Louis Pradel Hospital (Hospices Civils de Lyon, Lyon). The results of VO2peak predicted by the self-questionnaire will be compared to the VO2 peak measured during the examination.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* Patients considered stable according to the judgment of the investigator
* Indication of a stress test with measurement of VO2max as part of its medical management

Exclusion Criteria:

* Acute clinical event in the last 3 months
* System Illness Context
* Absence of coverage by a social security system
* Safeguarding justice (tutelage, guardianship, deprivation of civil rights)
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All stable patients above 18 years, referred for a VO2 peak test as part of their standard management in the Louis Pradel Hospital (Hospices Civils de Lyon, Lyon) and without acute clinical event in the last 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Capacity of the DASI self-questionnaire | Day 0
  Sensitivity and specificity of the DASI self-questionnaire translated into French to identify patients with a threshold of VO2max <14 milliliters (mL) O2 kilogram-1 minute-1 measured during the exercise test.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital louis Pradel, Bron, France